CLINICAL TRIAL: NCT02947542
Title: Use of Different Diagnostic Coronary Catheters Over the Radial Access - the UDDC - Radial Trial
Acronym: UDDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, David Manuel Leistner, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1.1
Record Dates: First submitted 2016-10-18; First posted 2016-10-28 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Stable Coronary Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BLK catheter (Experimental): Coronary angiography will be performed with the BLK catheter (one-catheter concept).
  Interventions: Device: One-catheter concept
- Tiger catheter (Experimental): Coronary angiography will be performed with the Tiger catheter (one-catheter concept).
  Interventions: Device: One-catheter concept
- Judkins catheter (Active Comparator): Coronary angiography will be performed with the Judkins catheter (standard catheter).
  Interventions: Device: Standard catheter

INTERVENTIONS:
Device: One-catheter concept — Coronary angiography will be performed using the one-catheter concept.
  Arms: BLK catheter; Tiger catheter
Device: Standard catheter — Coronary angiography will be performed using a standard catheter.
  Arms: Judkins catheter

SUMMARY:
There is no evidence from prospective randomized clinical trials regarding the performance of conventional (two-catheter-concept; TCC) versus one-catheter-concepts (OCC) for invasive coronary angiography over the radial access.

The aim of the present trial is to evaluate the efficacy and safety of different one-catheter concepts by use of the BLK and Tiger catheter compared to a TCC using standard Judkins catheters in diagnostic coronary angiography via transradial access. Patients with stable angina pectoris will be randomly assigned to coronary angiography performed with the BLK or Tiger (OCC) or Judkins catheters (TCC). The primary endpoint is coronary angiography duration.

DETAILED DESCRIPTION:
The aim of the present trial is to evaluate the efficacy and safety of a one-catheter concept using the BLK (Terumo, Somerset, USA) or the Tiger catheter (Terumo, Somerset, USA) compared to the standard Judkins catheters in diagnostic coronary angiography by the transradial access. Patients with stable angina pectoris will be randomly assigned to coronary angiography performed with the BLK (Group I), Tiger (Group II) or Judkins catheters (Group III). Primary endpoint is the time duration (sec) that is necessary to perform complete coronary angiography including 6 different projections for the left-coronary system and 3 different projections of the right-coronary-system. Secondary endpoints will cover safety and imaging quality of the different catheter systems.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 95 years
* Body weight > 60kg

Exclusion Criteria:

* Acute coronary syndrome or cardiogenic shock
* Contraindications for transracial access such as absence of radial pulse or abnormal Allen test
* Prior unsuccessful transradial coronary angiography
* Estimated glomerular filtration rate <40 ml/kg/min
* Patients not able to give informed consent
* Participation in another trial

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Coronary angiography Duration (sec) | Day 0 (corresponding to time point of procedure)
  assessed by Intention-to-treat analysis (IIT)

SECONDARY OUTCOMES:
Cross over rate to another catheter or transfemoral access. | Day 0 (corresponding to time point of procedure)
Flouroscopy time (sec) | Day 0 (corresponding to time point of procedure)
Contrast volume (ml) | Day 0 (corresponding to time point of procedure)
Safety endpoints (kinking, radial spasm, vascular access complications, bleeding complications). | Day 0 (corresponding to time point of procedure)
Imaging Quality (ostial stability, diagnostic value) | Day 0 (corresponding to time point of procedure)

CONTACTS AND LOCATIONS:
Overall Officials: David M Leistner, PD, Principal Investigator — Department of Cardiology, Campus Benjamin Franklin, Charité - Universitätsmedizin Berlin
Locations (1):
- Department of Cardiology, Campus Benjamin Franklin, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided